CLINICAL TRIAL: NCT01290432
Title: The Potential Effects of Inofolic Plus on Abnormal Ovarian Reserve Parameters in Subfertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palm Beach Center for Reproductive Medicine (Other)
Collaborators: Lo.Li. Pharma, Ltd. (Unknown)
Responsible Party: Principal Investigator, Scott Roseff, MD, Principal Investigator, Palm Beach Center for Reproductive Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Roseff-01
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Infertility, Female
Keywords: female fertility; ovarian reserve; oocyte quality; oocyte quantity; antimullerian hormone; AMH; dietary supplements; inofolic plus; myoinositol; folic acid
MeSH Terms: conditions — Infertility, Female | interventions — Folic Acid; Inositol; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inofolic Plus (Experimental): Patients are given Inofolic Plus to see if the AMH changes over a period of up to 90 days.
  Interventions: Dietary Supplement: Inofolic Plus

INTERVENTIONS:
Dietary Supplement: Inofolic Plus — Inofolic Plus contains folic acid and myoinositol and melatonin
  Other Names: folic acid, myoinositol, and melatonin in combination

SUMMARY:
Dr. Roseff and his colleagues are conducting a study to evaluate the effectiveness of a novel substance (Inofolic Plus®) in improving oocyte (egg) parameters in subfertile female patients, as measured through Anti-Mullerian Hormone (AMH) blood levels.

DETAILED DESCRIPTION:
Inofolic Plus® contains several nutritional elements including myo-inositol, melatonin, and folic acid. Myo-inositol was found to be helpful in improving egg quality and/or quantity in women with an ovarian abnormality called polycystic ovarian syndrome as well as in women without the disorder undergoing assisted reproduction.

Myo-inositol and folic acid are compounds that belong to the family of B-vitamins. Inositol is normally found in several types of foods. Folic acid has been found to significantly decrease the incidence of certain types of birth defects in women taking sufficient amounts prior to and during pregnancy. Preliminary studies using myo-inositol and folic acid demonstrated improvement in egg quality in-vitro and in-vivo as well as multiple metabolic parameters in women with irregular menstrual cycles and certain types of hormone imbalances.

Melatonin is a potent antioxidant. Folic acid is not classified as an antioxidant but has been reported to have antioxidant-like activity. Antioxidants have been given to infertile men for years to improve egg parameters. Most recently, studies have documented the efficacy of antioxidant treatment on human egg parameters and fertilization rates, especially in the setting of in-vitro fertilization (IVF). Inofolic Plus® contains melatonin and folic acid. Dr. Roseff hypothesizes that Inofolic Plus® may be effective in correcting abnormal egg parameters in women. A woman may have abnormal eggs from being exposed to environmental and workplace toxins that generate oxygen free radicals in her body (known as reactive oxygen species, or ROS). These ROS circulate through the blood stream and can enter the ovaries where eggs are stored. Eggs may be sensitive to ROS, and damage from the ROS may result in poor egg quality or quantity or both. The combination of nutrients and antioxidants in Inofolic Plus® may help to correct these abnormalities. Melatonin is a natural hormone normally found in the brain. This hormone helps regulate sleep/wake cycles. Melatonin levels increase during the evening and remain high during the night. This elevated level of melatonin is thought to induce drowsiness. It is because of this effect that we recommend taking Inofolic Plus® in the late evening near bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 - 42 years of age
* Diagnosed with "Diminished Ovarian Reserve" (DOR)

Exclusion Criteria:

* Ongoing history of illicit drug or tobacco use
* Ovarian surgery within 90 days of signing the consent form

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Potential Effects of Inofolic Plus on Abnormal Ovarian Reserve (AMH Levels) | Three Months
  Women will receive Infolic Plus nightly for up to 90 days. Baseline AMH blood levels will be analyzed, and AMH titers will be checked monthly thereafter for the 90 day duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Roseff, MD, Principal Investigator — Palm Beach Center for Reproductive Medicine
Locations (1):
- Palm Beach Center for Reproductive Medicine, Wellington, Florida, United States

REFERENCES:
- [Background] Tamura H, Takasaki A, Miwa I, Taniguchi K, Maekawa R, Asada H, Taketani T, Matsuoka A, Yamagata Y, Shimamura K, Morioka H, Ishikawa H, Reiter RJ, Sugino N. Oxidative stress impairs oocyte quality and melatonin protects oocytes from free radical damage and improves fertilization rate. J Pineal Res. 2008 Apr;44(3):280-7. doi: 10.1111/j.1600-079X.2007.00524.x. PMID 18339123
- [Background] Tamura H, Nakamura Y, Korkmaz A, Manchester LC, Tan DX, Sugino N, Reiter RJ. Melatonin and the ovary: physiological and pathophysiological implications. Fertil Steril. 2009 Jul;92(1):328-43. doi: 10.1016/j.fertnstert.2008.05.016. Epub 2008 Sep 18. PMID 18804205
- [Background] Papaleo E, Unfer V, Baillargeon JP, Fusi F, Occhi F, De Santis L. RETRACTED: Myo-inositol may improve oocyte quality in intracytoplasmic sperm injection cycles. A prospective, controlled, randomized trial. Fertil Steril. 2009 May;91(5):1750-1754. doi: 10.1016/j.fertnstert.2008.01.088. Epub 2008 May 7. PMID 18462730
- [Background] Papaleo E, Unfer V, Baillargeon JP, Chiu TT. Contribution of myo-inositol to reproduction. Eur J Obstet Gynecol Reprod Biol. 2009 Dec;147(2):120-3. doi: 10.1016/j.ejogrb.2009.09.008. Epub 2009 Oct 2. PMID 19800728